CLINICAL TRIAL: NCT01806324
Title: A Study to Evaluate Pharmacokinetics and Potential Drug Interactions of a Fixed-dose Combination Tablet, HL-040XC, in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HL-040XC-US-001
Record Dates: First submitted 2012-04-18; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Losartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HL040XC(Atorvastatin+Losartan) (Experimental): HL040XC lag time released combination drug
  Interventions: Drug: HL040XC
- Losartan + Atorvastatin (Active Comparator): Coadministration group
  Interventions: Drug: Losartan + Atorvastatin

INTERVENTIONS:
Drug: HL040XC — single dose
  Arms: HL040XC(Atorvastatin+Losartan)
Drug: Losartan + Atorvastatin — Single dose
  Arms: Losartan + Atorvastatin

SUMMARY:
The objective of this study is:

To evaluate the pharmacokinetics and safety of an experimental combination tablet containing 20 mg atorvastatin and 50 mg losartan potassium when administered orally as a single dose to healthy male subjects, compared with the concomitant administration of 20 mg atorvastatin and 50 mg losartan potassium tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 19 and 50 years of age, inclusive.
2. Subjects who weigh at least 121 pounds (55 kg), and are within ± 20% of their of ideal body weight (IBW). IBW (kg) = [height (cm) - 100] x 0.9.
3. Subjects who don't have any congenital or chronic disease.
4. Subjects who don't have any clinically significant abnormality on vital sign measurement, physical examination, clinical lab test, and ECG test at Screening.
5. Subjects who are able to read and understand the consent form.

Exclusion Criteria:

1. Subjects who have any history or presence of hypersensitivity to HMG-CoA reductase inhibitors such as atorvastatin or angiotensin receptor blockers such as losartan.
2. Subjects who have any medical history that may affect the absorption, distribution, metabolism, and excretion of study drugs (e.g., cardiovascular, respiratory, renal, endocrinal, hematological, digestive, neurological, or psychiatric disease).
3. Subjects who have a creatinine clearance < 80 mL/min, which is calculated by Cockcroft-Gault equation: (140 - age) x (Wt in kg) / (72 x sCr).
4. Subjects who had a severe injury or surgery within 4 weeks prior to Screening.
5. Subjects who have a positive drug screen.
6. Subjects who take any prescription or herbal drug within 1 week prior to Screening.
7. Subjects who take any over-the counter (OTC) drug, which may affect this study or the subject's safety according to the judgment of investigator, at Screening.
8. Subjects who take any herbal drug containing St. John's Wort or other drugs, which are metabolized by CYP3A4 enzyme or inhibit or stimulate CYP enzyme (e.g., itraconazole, ketoconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitor, nefazodone) within 4 weeks prior to Screening.
9. Subjects who have abnormal meal pattern that may affect the absorption, distribution, metabolism, and excretion of study drugs (e.g., taking grapefruit juice over 1 L per day).
10. Subjects who received an investigational product within 4 weeks prior to Screening.
11. Subjects who have donated blood within 6 weeks prior to Screening.
12. Subjects who consume alcohol over 21 units per week (1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol) and can't accept the prohibition of alcohol during this clinical study.
13. Subjects who smoke more than 10 cigarettes per day.
14. Subjects who have low blood pressure (systolic ≤ 100 mmHg or diastolic ≤ 65 mmHg) or high blood pressure (systolic ≥ 150 mmHg or diastolic ≥ 95 mmHg) at Screening.
15. Subjects who test positive on serology HBsAg, HCV Ab, HIV Ab or VDRL at Screening.
16. Subjects who have active liver disease or elevated serum transaminase level higher than 3 times of upper limit of normal.
17. Subjects who have the inability in the opinion of the investigator to comply with the protocol.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 ~ 48hr
  To evaluate its bioequivalency in Cmax and AUC of each test group
AUC | 0~48HR
  To evaluate bioequvalency of each group

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States